CLINICAL TRIAL: NCT06788912
Title: KEYMAKER-U01 Substudy 01E: A Phase 2 Umbrella Study With Rolling Arms of Investigational Agents With or Without Chemotherapy in Combination With Pembrolizumab in Treatment of Participants With Newly Diagnosed Resectable Stages II-IIIB (N2) Non-small Cell Lung Cancer (NSCLC)
Brief Title: Pembrolizumab (MK-3475) Plus Investigational Agents in Resectable Non-small Cell Lung Cancer (NSCLC) (MK-3475-01E/KEYMAKER-U01)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3475-01E; MK-3475-01E (Other: MSD Protocol Number); KEYMAKER-U01 (Other: MSD); 2023-509234-19-00 (Registry Identifier: EU CT); U1111-1299-6753 (Registry Identifier: UTN)
Record Dates: First submitted 2025-01-17; First posted 2025-01-23 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Lung Neoplasm Malignant
Keywords: Programmed Cell Death-1 (PD1, PD-1); Programmed Cell Death 1 Ligand 1(PDL1, PD-L1); Programmed Cell Death 1 Ligand 2 (PDL2, PD-L2)
MeSH Terms: conditions — Lung Neoplasms; Parkinson Disease 4, Autosomal Dominant Lewy Body | interventions — pembrolizumab; Neoadjuvant Therapy; Cisplatin; Gemcitabine; Pemetrexed; Histamine Antagonists; Histamine H2 Antagonists; Acetaminophen; Dexamethasone; Carboplatin; Adjuvants, Pharmaceutic; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Pembrolizumab + Platinum (Active Comparator): Neoadjuvant: Prior to surgery pembrolizumab 200 mg every three weeks (Q3W) for 4 cycles (each cycle is 21 days); Cisplatin 75 mg/m^2 Q3W with gemcitabine 1000 mg/m^2 on Day 1 and Day 8 Q3W (squamous tumors), pemetrexed 500 mg/m^2 Q3W (nonsquamous tumors), or paclitaxel 175 mg/m^2 or 200 mg/m^2 q3w (any histology) OR Carboplatin AUC 5 mg/mL• min or AUC 6 mg/mL• min with paclitaxel 175 mg/m^2 or 200 mg/m^2 Q3W (any histology), pemetrexed 500 mg/m^2 Q3W (nonsquamous tumors), or gemcitabine 1000 mg/m^2 on Day 1 and Day 8 Q3W (squamous tumors); followed by surgery.
  Adjuvant: After surgery pembrolizumab 200 mg Q3W for 13 cycles (each cycle is 21 days).
  Interventions: Biological: Pembrolizumab (neoadjuvant); Drug: Cisplatin; Drug: Gemcitabine; Drug: Pemetrexed; Drug: Carboplatin; Biological: Pembrolizumab (adjuvant); Drug: Paclitaxel
- Pembrolizumab + Sacituzumab tirumotecan (Experimental): Neoadjuvant: Prior to surgery pembrolizumab 200 mg Q3W for 4 cycles (each cycle is 21 days); sacituzumab tirumotecan 4 mg/kg Q2W for 6 cycles (each cycle is 14 days), followed by surgery.
  Adjuvant: After surgery pembrolizumab 200 mg Q3W for 13 cycles (each cycle is 21 days). Optional adjuvant platinum-based doublet chemotherapy up to 4 cycles may be given at the investigator's discretion.
  Interventions: Biological: Pembrolizumab (neoadjuvant); Drug: Cisplatin; Drug: Gemcitabine; Drug: Pemetrexed; Drug: Sacituzumab tirumotecan; Drug: H1 receptor antagonist; Drug: H2 receptor antagonist; Drug: Acetaminophen (or equivalent); Drug: Dexamethasone (or equivalent); Drug: Carboplatin; Biological: Pembrolizumab (adjuvant); Drug: Paclitaxel; Drug: Steroid mouthwash (dexamethasone or equivalent)

INTERVENTIONS:
Biological: Pembrolizumab (neoadjuvant) — Before surgery neoadjuvant Pembrolizumab 200 mg by intravenous (IV) infusion on day 1 of each 21-day cycle for 4 cycles
  Other Names: KEYTRUDA®; MK-3475
Drug: Cisplatin — Cisplatin 75 mg/m^2 by IV infusion on day 1 of each 21-day cycle for 4 cycles
  Other Names: PLATINOL®
Drug: Gemcitabine — In squamous tumors Gemcitabine 1000 mg/m^2 by IV infusion on day 1 and day 8 of each 21-day cycle for 4 cycles.
  Other Names: GEMZAR®
Drug: Pemetrexed — In nonsquamous tumors Pemetrexed 500 mg/m^2 by IV infusion on day 1 of each 21-day cycle for 4 cycles
  Other Names: Alimta®
Drug: Sacituzumab tirumotecan — Sacituzumab tirumotecan 4 mg/kg by IV infusion on day 1 of each 14-day cycle for up to 6 cycles
  Other Names: MK-2870; SKB264
  Arms: Pembrolizumab + Sacituzumab tirumotecan
Drug: H1 receptor antagonist — Administered as rescue medication before Sacituzumab tirumotecan infusion per approved product label
  Arms: Pembrolizumab + Sacituzumab tirumotecan
Drug: H2 receptor antagonist — Administered as rescue medication before Sacituzumab tirumotecan infusion per approved product label
  Arms: Pembrolizumab + Sacituzumab tirumotecan
Drug: Acetaminophen (or equivalent) — Administered as rescue medication before Sacituzumab tirumotecan infusion per approved product label
  Arms: Pembrolizumab + Sacituzumab tirumotecan
Drug: Dexamethasone (or equivalent) — Administered as rescue medication 8 -10 mg before Sacituzumab tirumotecan infusion per approved product label
  Arms: Pembrolizumab + Sacituzumab tirumotecan
Drug: Carboplatin — AUC 5 mg/mL min or AUC 6 mg/mL min by IV infusion on day 1 of each 21-day cycle for 4 cycles
  Other Names: PARAPLATIN®
Biological: Pembrolizumab (adjuvant) — After surgery adjuvant Pembrolizumab 200 mg by IV infusion on day 1 of each 21-day cycle for 13 cycles
  Other Names: KEYTRUDA®; MK-3475
Drug: Paclitaxel — Paclitaxel 175 or 200 mg/m^2 by IV infusion on day 1 of each 21-day cycle for 4 cycles.
Drug: Steroid mouthwash (dexamethasone or equivalent) — Administered orally as rescue medication 2-5 mL 4 times daily
  Arms: Pembrolizumab + Sacituzumab tirumotecan

SUMMARY:
The main goals are after treatment given before surgery, to measure the number of people who have no signs of cancer cells in tumors and lymph nodes removed during surgery; and to learn about whether the cancer gets smaller or goes away by measuring the number of people with a certain number of living cancer cells in the tumor removed during surgery.

ELIGIBILITY:
The main inclusion and exclusion criteria include but are not limited to the following:

Inclusion Criteria:

* Has previously untreated and pathologically confirmed resectable Stage II, IIIA, or IIIB (N2) non-small cell lung cancer (NSCLC)
* Able to undergo protocol therapy, including necessary surgery
* Confirmation that epidermal growth factor receptor (EGFR) -directed therapy is not indicated as primary therapy
* Has an Eastern Cooperative Oncology Group (ECOG) performance status of either 0 or 1 as assessed within 10 days before initiation of study intervention.
* Is able to provide archival or newly obtained core/excisional biopsy of the primary lung tumor or lymph node metastasis.

Exclusion Criteria:

* Has one of the following tumor locations/types: NSCLC involving the superior sulcus, large-cell neuro-endocrine cancer, mixed tumors containing small cell and non-small cell elements, or sarcomatoid tumor.
* Has Grade ≥2 peripheral neuropathy.
* Has history of documented severe dry eye syndrome, severe Meibomian gland disease and/or blepharitis, or severe corneal disease that prevents/delays corneal healing.
* Has active inflammatory bowel disease requiring immunosuppressive medication or previous history of inflammatory bowel disease (eg, Crohn's disease, ulcerative colitis, or chronic diarrhea).
* Has uncontrolled, significant cardiovascular disease or cerebrovascular disease.
* Received a live or live-attenuated vaccine within 30 days before the first dose of study intervention
* Received prior radiotherapy within 2 weeks of start of study intervention, or radiation related toxicities, requiring corticosteroids.
* Diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study intervention.
* Known additional malignancy that is progressing or has required active treatment within the past 5 years.
* Severe hypersensitivity (≥Grade 3) to pembrolizumab and/or any of its excipients.
* Active autoimmune disease that has required systemic treatment in the past 2 years. Replacement therapy (e.g. thyroxine, insulin, or physiologic corticosteroid) is allowed.
* History of (noninfectious) pneumonitis/interstitial lung disease that required steroids or has current pneumonitis/interstitial lung disease.
* Active infection requiring systemic therapy.
* Hepatitis B (defined as hepatitis B surface antigen [HBsAg] reactive) or Hepatitis C virus (defined as detectable hepatitis C virus (HCV) ribonucleic acid (RNA) [qualitative]) infection.
* Known history of human immunodeficiency virus (HIV) infection.
* History of allogeneic tissue/solid organ transplant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-03-20 (Actual); Primary Completion 2032-02-06 (Estimated); Study Completion 2032-02-06 (Estimated)

PRIMARY OUTCOMES:
Pathological Complete Response (pCR) | Up to approximately 20 weeks
  pCR is defined as absence of residual viable invasive cancer on hematoxylin- and eosin-stained slides of the resected lung specimen and lymph nodes.
Percent Residual Viable Tumor (%RVT) | Up to approximately 20 weeks
  %RVT is defined as the percentage of residual tumor estimated by comparing the estimated cross-sectional area of viable tumor with estimated cross-sectional areas of remainder of tumor bed. The tumor bed is defined as the area of tissue occupied by viable tumor or tumoral regression (includes areas of necrosis, foamy macrophages, giant cell reaction, cholesterol cleft granuloma, and inflammation.)

SECONDARY OUTCOMES:
Percentage of Participants Who Report at Least 1 Adverse Event (AE) | Up to approximately 5 years
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study intervention.
Percentage of Participants Who Discontinue Study Treatment Due to an AE | Up to approximately 1 year
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study intervention.
Event-free Survival (EFS) | Up to approximately 5 years
  EFS is defined as the time from randomization to any of the following events: radiographic disease progression per Response Evaluation Criteria In Solid Tumors 1.1 (RECIST 1.1) (for participants who have not had or will not have surgery, or participants who have gross residual disease after an incomplete resection [R2 resection]); local progression (primary tumor or regional lymph nodes) or distant metastasis precluding planned surgery; tumor determined to be unresectable in the operating room; local or distant recurrence (for participants who are disease free after surgery or participants with microscopic positive margins [R1 resection]); occurrence of new primary NCSLC; death due to any cause.
Overall Survival (OS) | Up to approximately 5 years
  OS is defined as the time from randomization to death due to any cause.
Distant Metastasis-Free Survival (DMFS) | Up to approximately 5 years
  DMFS is defined as the time from randomization to the date of diagnosis of distant metastasis or death, whichever occurs first.
Objective Response Rate (ORR) | Up to approximately 12 weeks
  OR is defined as a complete response or partial response with or without confirmation per RECIST 1.1 as assessed by the investigator during the Neoadjuvant Phase.
Percentage of Participants Who Experience a Perioperative Complication | Up to approximately 20 weeks
  Perioperative Complications include both intraoperative and postoperative complications.
Mean Length of Hospital Stay | Up to approximately 20 weeks
  Hospital Stay is the length of inpatient time spent in hospital.
Percentage of Participants Who Require Hospital Readmission after Discharge | Up to approximately 20 weeks
  In participants previously discharged from hospital, the percentage requiring readmission to hospital.
Mean Length of Surgery | Up to approximately 20 weeks
  Length of surgery is the time spent in surgery.
Percentage of Participants Who Require a Blood Transfusion | Up to approximately 20 weeks
  Blood transfusion is the transfer of donated blood into the vein of a recipient.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (28):
- United States (2):
  - Sansum Clinic (Ridley Tree) ( Site 8012), Santa Barbara, California
  - MedStar Franklin Square Medical Center ( Site 0033), Baltimore, Maryland
- Chile (3):
  - Centro de Estudios Clínicos SAGA ( Site 0162), Santiago, Region M. de Santiago
  - FALP ( Site 0161), Santiago, Region M. de Santiago
  - Bradfordhill ( Site 0160), Santiago, Region M. de Santiago
- Greece (4):
  - Alexandra General Hospital of Athens Oncology-Hematology Unit ( Site 0203), Athens, Attica
  - ATTIKON GENERAL UNIVERSITY HOSPITAL-Oncology ( Site 0202), Athens, Attica
  - Metropolitan Hospital-4th Oncology Dept ( Site 0201), Athens, Attica
  - University General Hospital of Heraklion ( Site 0200), Heraklion, Irakleio
- Hungary (3):
  - Petz Aladar Egyetemi Oktato Korhaz-Pulmonológia (Dr. Szalai Zsuzsanna) ( Site 0062), Győr, Győr-Moson-Sopron
  - Jász-Nagykun-Szolnok Vármegyei Hetényi Géza Kórház-Onkologiai Kozpont ( Site 0061), Szolnok, Jász-Nagykun-Szolnok
  - Országos Korányi Pulmonológiai Intézet ( Site 0060), Budapest
- Italy (4):
  - Azienda Ospedaliera Universitaria Careggi ( Site 0173), Florence, Tuscany
  - Ospedale San Raffaele. ( Site 0171), Milan
  - Fondazione IRCCS Istituto Nazionale dei Tumori ( Site 0175), Milan
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS - Università Cattolica del Sacro Cuore ( Site 0174), Roma
- Poland (3):
  - Wielkopolskie Centrum Pulmonologii i Torakochirurgii-Oddzial Onkologii Klinicznej z Pododdzialem Dz ( Site 0153), Poznan, Greater Poland Voivodeship
  - Narodowy Instytut Onkologii im. Marii Sklodowskiej-Curie - P-Klinika Nowotworow Pluca i Klatki Pier ( Site 0151), Warsaw, Masovian Voivodeship
  - Uniwersyteckie Centrum Kliniczne-Early Clinical Trials Unit ( Site 0150), Gdansk, Pomeranian Voivodeship
- Hospital Clínic de Barcelona ( Site 0092), Barcelona, Spain
- Hacettepe Universite Hastaneleri-oncology hospital ( Site 0700), Ankara, Turkey (Türkiye)
- Ukraine (7):
  - CNE CC of Oncology Hematol ( Site 0130), Cherkasy, Cherkasy Oblast
  - Municipal Enterprise "Bukovinian сlinical oncology сenter" ( Site 0139), Chernivtsi, Chernivetska Oblast
  - CNCE Precarpathian Clinical Oncologic Center ( Site 0131), Ivano-Frankivsk, Ivano-Frankivsk Oblast
  - MNPE LTMU Multidisc. Clin. Hosp. of Emerg. and Intens. Care ( Site 0132), Lviv, Lviv Oblast
  - ME RIVNE REGIONAL ANTITUMOR CENTER ( Site 0460), Rivne, Rivne Oblast
  - Communal Noncommercial Enterprise "Podillia Regional Oncology Center Of Vinnytsia Regional Council" ( Site 0135), Vinnytsia, Vinnytsia Oblast
  - Shalimov Institute of Surgery and Transplantation ( Site 0138), Kyiv

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/